CLINICAL TRIAL: NCT05114746
Title: A Prospective, Open Label, Multicenter, Single Arm, Phase 2 Study of 177Lu-PSMA-617 in the Treatment of Participants With Progressive PSMA- Positive Metastatic Castration-resistant Prostate Cancer (mCRPC) in Japan
Brief Title: Study of 177Lu-PSMA-617 In Metastatic Castrate-Resistant Prostate Cancer in Japan
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Eckert & Ziegler Radiopharma GmbH (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA617A11201
Record Dates: First submitted 2021-09-29; First posted 2021-11-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: 177Lu-PSMA-617; 68Ga-PSMA-11; 68Ge/68Ga Generator; metastatic castration-resistant prostate cancer; mCRPC; prostate-specific membrane antigen; PSMA; radioligand; taxane; enzalutamide; abiraterone; Overall Response Rate; ORR
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-PSMA-617 (Experimental): PSMA positivity will be confirmed by PET/CT scan after administration of 68Ga-PSMA-11. All eligible participants will receive recommended dose of 177Lu-PSMA-617 via intravenous injection every 6 weeks (+/- 1 week) for a maximum of 6 cycles.
  Interventions: Radiation: 177Lu-PSMA-617; Radiation: 68Ga-PSMA-11; Other: Best supportive/best standard of care

INTERVENTIONS:
Radiation: 177Lu-PSMA-617 — administered intravenously at a dose of 7.4 GBq (+/- 10%). 7.4 GBq dose is equivalent to 200 mCi or 7400 MBq.
Radiation: 68Ga-PSMA-11 — 68Ga-PSMA-11 is manufactured by radiolabeling of PSMA-11 precursor with 68Ga directly at clinical trial sites immediately prior to administration into participants. The 68Ga used for radiolabeling will be eluted from the 68Ge/68Ga generator. 68Ga-PSMA-11 will be prepared as a sterile solution and administered intravenously at a dose of 111 - 259 MBq (3 - 7 mCi).
Other: Best supportive/best standard of care — Best supportive/best standard of care as defined by the local investigator (Post taxane population only)

SUMMARY:
The purpose of this study is to assess the efficacy, tolerability, safety, pharmacokinetic (PK) and dosimetry of 177Lu-PSMA-617, in participants with progressive prostate-specific membrane antigen (PSMA)-positive metastatic castration-resistant prostate cancer (mCRPC) in Japan. Furthermore, the safety, PK and dosimetry of 68Ga-PSMA-11 (PSMA imaging agent) are assessed in the same study.

Another purpose of this study is to provide humanistic perspective access to study treatment (68Ga-PSMA-11 and 177Lu-PSMA-617) for the eligible patients with PSMA-positive mCRPC until marketed products are available in Japan.

Furthermore, if data availability PK and dose rate of 177 Lu-PSMA-617 will be evaluated to refine discharge criteria in Japan.

After obtaining manufacturing and marketing approval in Japan, this clinical trial will continue as a post marketing trial.

DETAILED DESCRIPTION:
This study is an open label, multicenter, single arm, phase II study to evaluate the efficacy, tolerability, safety, PK and dosimetry of 177Lu-PSMA-617 in participants with progressive PSMA-positive mCRPC in Japan. Furthermore, the safety, PK, and dosimetry of 68Ga-PSMA-11 (PSMA imaging agent) are also evaluated in this study.

This study consists of two populations:

1. Post-taxane population:

   The post-taxane population will include men with PSMA-positive mCRPC who received at least one ARDT (for example enzalutamide, abiraterone etc.) and were previously treated with at least one, but no more than two taxane regimens. Participants treated with only 1 prior taxane regimen are eligible if the participant's physician deems the participants unsuitable to receive a second taxane regimen.
2. Pre-taxane population; The pre-taxane population will include men with PSMA-positive mCRPC who were previously treated with one ARDT as last treatment and have not been exposed to a taxane-containing regimen in the CRPC or HSPC settings and for whom it is considered appropriate to delay taxane-based chemotherapy.

This is a 4-part study: Part 1 (a safety run-in part), Part 2 (post-taxane part), Part 3 (pre-taxane part) and Part 4 (expanded trial part).

1. Part 1 (safety run-in part) will confirm the tolerability and safety of recommended regimen, once every 6-weeks, 7.4 GBq of the 177Lu-PSMA-617. Minimum of 3 participants as 177Lu-PSMA-617 tolerability evaluable participants will be enrolled. Dosimetry and PK assessments of 177Lu-PSMA-617 are mandatory for participants enrolled in this part.
2. Part 2 (post-taxane part) will evaluate the efficacy, safety, PK and dosimetry of 177Lu-PSMA-617 plus BSC/BSoC, as well as safety, PK, and dosimetry of 68Ga-PSMA-11 in post-taxane participants with PSMA-positive mCRPC.
3. Part 3 (pre-taxane part) will evaluate the efficacy, safety, PK and dosimetry of 177Lu-PSMA-617, as well as safety, PK, and dosimetry of 68Ga-PSMA-11 in taxane naïve participants with PSMA-positive mCRPC
4. Part 4 (expanded trial part) will provide humanistic perspective access of study treatment (68Ga-PSMA-11 and 177Lu-PSMA-617) for the Japanese post-taxane participants with PSMA-positive mCRPC until marketed products are available in Japan. Additional safety and efficacy of 68Ga-PSMA-11 and of 177Lu-PSMA-617 will be evaluated.

Additionally, PK and dose rate will be evaluated (PK is optional and dose rate is mandatory in Part 4).

Approximately 80 eligible participants will be enrolled in Part 4 and approximately 10 evaluable participants PK data will be collected.

This study will consist of 3 periods: screening period, treatment period, and long term follow up.

The long-term follow-up ends after participant transitions to a post marketing trial.

ELIGIBILITY:
Key Inclusion Criteria:

* ECOG performance status:

  1. Post-taxane population only: 0 to 2.
  2. Pre-taxane population only: 0 to 1.
* Participants must have a previous histological, pathological, and/or cytological confirmation of prostate cancer.
* Part 1/2/3 only; Participants must have a positive 68Ga-PSMA-11 PET/CT scan, as determined by the sponsor's central reader, before the enrollment to 177Lu-PSMA-617 treatment period.
* Participants must have a positive 68Ga-PSMA-11 PET/CT scan, as determined by the local investigator, before the enrollment to 177Lu-PSMA-617 treatment period.
* Participants must have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L).
* Post-taxane population only: Participants must have received at least one ARDT (for example enzalutamide, abiraterone, apalutamide, or darolutamide, etc.) in either the hormone-sensitive/castrate-resistant or non-metastatic/metastatic prostate cancer setting.
* Pre-taxane population only: Participants must have progressed only once on prior second generation ARDT (abiraterone, enzalutamide, darolutamide, or apalutamide) and be a candidate for change in ARDT as assessed by the treating physician.

  1. first generation androgen receptor inhibitor therapy (e.g. bicalutamide) is allowed but not considered as prior ARDT therapy
  2. second generation ARDT must be the most recent therapy received.
* Post-taxane population only: Participants must have been previously treated with at least 1, but no more than 2 prior taxane regimens. A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. If a participant has received only 1 taxane regimen, the participant is eligible if :

  a. The participant's physician deems him unsuitable to receive a second taxane regimen (e.g., frailty assessed by geriatric or health status evaluation or intolerance, etc.).
* Participants must have progressive mCRPC. Documented progressive mCRPC will be based on at least 1 of the following criteria:

  1. Serum PSA progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. 1.0 ng/mL is the minimal starting value if confirmed rise in PSA is the only indication of progression.
  2. Soft-tissue progression defined as an increase >= 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions.
  3. Progression of bone disease: two new lesions; only positivity on the bone scan defines metastatic disease to bone (PCWG3 criteria, Scher et al 2016).
* Part 1/2/3 only; Participants must have at least one measurable lesion per PCWG3-modified RECIST v1.1 on CT or MRI.

Key Exclusion Criteria:

* Previous treatment with any of the following within 6 months of the enrollment: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation. Previous PSMA-targeted therapy is not allowed.
* Post-taxane population: Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies], ARDT is not included) within 28 days prior to day of the enrollment.
* Pre-taxane population: Prior treatment with PARP inhibitor, cytotoxic chemotherapy for castration resistant or castrate sensitive prostate cancer (e.g., taxanes, platinum, estramustine, vincristine, methotrexate, etc.), immunotherapy or biological therapy [including monoclonal antibodies]) [Note: Taxane exposure (maximum 6 cycles) in the adjuvant or neoadjuvant setting is allowed if 12 months have elapsed since completion of this adjuvant or neoadjuvant therapy]
* Known hypersensitivity to the components of 177Lu-PSMA-617, 68Ga-PSMA-11 or excipients or to drugs of similar classes.
* Concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, PARP inhibitors, biological, AKT inhibitors or investigational therapy.
* Participants with a history of CNS metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity.
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.

Ages: 20 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 110 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 (safety run-in part): Dose Limiting Toxicity (DLT) during 1 cycle (6 weeks) | Cycle 2 Day 1 (Day 42)
  A Dose Limiting Toxicity (DLT) is defined as any toxicity not attributable to the disease or disease-related processes under investigation, the time window for DLT assessment period is Cycle 1. To be considered a DLT, it must be related to 177Lu-PSMA-617 while fulfilling one of the criteria as per the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Part 2 (Post-taxane part) and Part 3 (Pre-taxane part): Overall Response Rate (ORR) based on local assessment | From date of the first administration of 177Lu-PSMA-617 until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Overall Response Rate (ORR) is defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) according to PCWG3 modified RECIST 1.1.

SECONDARY OUTCOMES:
Part 2 and Part 3 (main part): Overall Survival (OS) | From date of the first administration of 177Lu-PSMA-617 until date of death from any cause, assessed up to 2 years
  Overall survival (OS) is defined as the time (in months) from the date of the first administration of 177Lu-PSMA-617 to the date of death due to any cause. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive (on or before the cut-off date).
Part 2 and Part 3 (main part): Radiographic Progression-Free-Survival (rPFS) based on local assessment | From date of the first administration of 177Lu-PSMA-617 until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Radiographic progression free survival (rPFS) is defined as the time (in months) from the date of the first administration of 177Lu-PSMA-617 to the date of radiographic progression as outlined in PCWG3 guideline or death due to any cause. The local radiographic imaging assessment will be used. In case, there are participants without measurable lesion at baseline based on local review per PCWG3-modified RECIST v1.1 in primary analysis set, rPFS will be assessed for participants with measurable disease, and for participants regardless of existing measurable disease as well.
Part 2 and Part 3 (main part): Overall Response Rate (ORR) based on central review | From date of the first administration of 177Lu-PSMA-617 until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Overall response rate (ORR) is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR), as per central review and according to PCWG3-modified RECIST v1.1. ORR will be assessed for participants who have evaluable disease by PCWG3-modified RECIST at baseline only.
Part 2 and Part 3 (main part): Disease Control Rate (DCR) as per central and local review | From date of the first administration of 177Lu-PSMA-617 until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Disease control rate (DCR) is defined as the proportion of participants with best overall response (BOR) of complete response (CR), partial response (PR) or stable disease (SD), as per central and local review and according to PCWG3-modified RECIST v1.1. DCR will be assess for participants who have evaluable disease by PCWG3-modified RECIST at baseline only.
Part 2 and Part 3 (main part): Duration of Response (DOR) based on local imaging | From the date of the first documented response (CR or PR) to the date of first documented progression or death due to any cause, assessed up to 2 years
  Duration of response (DOR) is defined as the time (in months) from the date of the first documented response (CR or PR) to the date of first documented progression according to PCWG3-modified RECIST v1.1 or death due to any cause, among participants with a confirmed response. The local imaging assessment will be used. DOR will be assessed for participants who have an evaluable disease by PCWG3-modified RECIST v1.1 at baseline only.
Part 2 and Part3 (main part): Time to first symptomatic skeletal event (SSE) of 177Lu-PSMA-617 | From the date of the first administration of 177Lu-PSMA-617 until the date of SSE or date of death from any cause, whichever comes first, assessed up to 2 years
  Time to a first symptomatic skeletal event (SSE) is defined as the time (in months) from the first administration of 177Lu-PSMA-617 to the date of SSE or death due to any cause. SSE date is date of the first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain, or death due to any cause, whichever comes first. SSE date for this endpoint is collected up through the end of treatment visit.
Part 2 and Part 3 (main part): Progression Free Survival (PFS) | From the date of the first administration of 177Lu-PSMA-617 until the date of progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Progression Free Survival (PFS) (Radiographic/clinical/PSA) is defined as the time (in months) from the date of the first administration of 177Lu-PSMA-617 to the date of radiographic, clinical or PSA progression free survival, or death due to any cause, whichever occurs first. The local radiographic imaging assessment will be used. In case, there are participants without measurable lesion at baseline based on local review per PCWG3-modified RECIST v1.1 in primary analysis set, PFS will be assessed for participants with a measurable disease, and for participants regardless of existing measurable disease as well.
Part 2 and Part 3 (main part): Percentage of Participants with Biochemical Response as measured by Prostate Specific Antigen (PSA) | From Baseline till 30 days safety follow-up, assessed up to 2 years
  PSA response rate is defined as the proportion of participants with PSA response that is defined as PSA decrease of >= 50% from baseline that is confirmed by a second consecutive PSA measurement >= 4 weeks later. Local laboratory assessments will be used. Determination of response status will be based on Prostate Cancer Working Group 3 (PCWG3) recommendations.
Part 2 and Part 3 (main part): Change from Baseline in European Quality of Life (EuroQol) - 5 Domain 5 Level scale (EQ-5D- 5L) | From Baseline up till end of treatment visit, an average of 13 months
  EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Part 2 and Part 3 (main part): Change from Baseline in Functional Assessment of Cancer Therapy - Prostate (FACT-P) Questionnaire | From Baseline up till end of treatment visit, an average of 13 months
  FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACTGeneral (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Part 2 and Part 3 (main part): Change from Baseline in Brief Pain Inventory - Short Form (BPISF) Questionnaire: Pain Severity Score | From Baseline up till end of treatment visit, an average of 13 months
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item selfreport questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain severity score is a mean value for BPI-SF questions 3, 4, 5 and 6 (questions inquiring about the extent of pain, where the extent is ranked from 0 [no pain] to 10 [pain as bad as you can imagine]). Pain severity progression is defined as an increase in score of 30% or greater from baseline without decrease in analgesic use.
Part 2 and Part 3 (main part): Change from Baseline in Brief Pain Inventory - Short Form (BPISF) Questionnaire: Pain Interference Score | From Baseline up till end of treatment visit, an average of 13 months
  The BPI-SF is a publicly available instrument to assess the pain and includes severity and interference scores. BPI-SF is an 11-item self report questionnaire that is designed to assess the severity and impact of pain on daily functions of a participant. Pain interference score is mean value for the 7 BPI-SF questions (questions inquiring about the extent of interference with activities by pain) where the extent is ranked from 0 (does not interfere) to 10 (completely interferes). Pain interference progression is defined as an increase in score of 50% or greater from baseline without decrease in analgesic use.
Part 2 and Part 3 (main part): Percentage of Participants with treatment emergent adverse events | From Baseline till 30 days safety follow-up, assessed up to 2 years
  Safety measured by the percentage of participants with treatment emergent adverse events (events started after the first dose of study medication or events present prior to start of treatment but increased in severity based on preferred term).
Part 2 and Part 3 (main part): Absorbed dose and Effective whole-body dose 68Ga-PSMA-11 | 68Ga-PSMA-11 PET imaging acquired at Day 1 (0, 20, 40 , 60, 90, 180 and 255 minutes post infusion)
  The absorbed dose in target organs and the effective radiation dose will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Part 2 and Part 3 (main part): Absorbed dose and Effective whole-body dose of 177Lu-PSMA-617 | 177Lu-PSMA-617 SPECT/CT imaging acquired at Day 1, 2, 3 and 8 of Cycle 1
  The absorbed dose in target organs and the effective radiation dose will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Part 2 and Part 3 (main part): Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main part): Time of maximum observed drug concentration occurrence (Tmax) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main part): Observed maximum plasma concentration (Cmax) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): Area Under the plasma concentration-time Curve from the time 0 to the last observed quantifiable concentration (AUC(0-t)) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t) will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): AUC(0-t) divided by the dose administered (AUC(0- t)/D) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t)/D will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): Terminal elimination half-life (T1/2) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-inf) will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): Total systemic clearance for intravenous administration (CL) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): volume of distribution during the terminal phase following intravenous elimination (Vz) of 68Ga-PSMA-11 | Cycle 1 Day 1 (0.083, 0.25, 0.5, 0.75, 1.42, 2.92 and 4.08 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main part): Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main part): Time of maximum observed drug concentration occurrence (Tmax) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main part): Observed maximum plasma concentration (Cmax) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): Area Under the plasma concentration-time Curve from the time 0 to the last observed quantifiable concentration (AUC(0-t)) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t) will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): AUC(0-t) divided by the dose administered (AUC(0- t)/D) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-t)/D will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): Terminal elimination half-life (T^1/2) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. The half-live will be listed and summarized using descriptive statistics
Part 2 and Part 3 (main study): Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC(0-inf) will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): Total systemic clearance for intravenous administration (CL) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL will be listed and summarized using descriptive statistics.
Part 2 and Part 3 (main study): volume of distribution during the terminal phase following intravenous elimination (Vz) of 177Lu-PSMA-617 | Cycle 1 Day 1 (0, 0.33, 1, 2 and 4 hours post infusion), Cycle 1 Day 2 (24 hours post infusion), Cycle 1 Day 3 (48 hours post infusion), Cycle 1 Day 4 (72 hours post infusion), Cycle 1 Day 6 (120 hours post infusion)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz will be listed and summarized using descriptive statistics.
Part 4 (expanded trial part): Overall Response Rate (ORR) based on local assessment | From date of the first administration of 177Lu-PSMA-617 until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Overall response rate (ORR) is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR), as per local investigator review and according to PCWG3-modified RECIST v1.1. ORR will be assessed for participants who have evaluable disease by PCWG3-modified RECIST at baseline only.
Part 4 (expanded trial part): Radiographic Progression-Free-Survival (rPFS) based on local assessment | From date of the first administration of 177Lu-PSMA-617 until date of radiographic progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Radiographic progression free survival (rPFS) is defined as the time (in months) from the date of the first administration of 177Lu-PSMA-617 to the date of radiographic progression as outlined in PCWG3 guideline or death due to any cause. The local radiographic imaging assessment will be used. In case, there are participants without measurable lesion at baseline based on local review per PCWG3-modified RECIST v1.1 in primary analysis set, rPFS will be assessed for participants with measurable disease, and for participants regardless of existing measurable disease as well.
Part 4 (expanded trial part): Progression Free Survival (PFS) | From the date of the first administration of 177Lu-PSMA-617 until the date of progression or date of death from any cause, whichever comes first, assessed up to 2 years
  Progression Free Survival (PFS) (Radiographic/clinical/PSA) is defined as the time (in months) from the date of the first administration of 177Lu-PSMA-617 to the date of radiographic, clinical or PSA progression free survival, or death due to any cause, whichever occurs first. The local radiographic imaging assessment will be used. In case, there are participants without measurable lesion at baseline based on local review per PCWG3-modified RECIST v1.1 in primary analysis set, PFS will be assessed for participants with a measurable disease, and for participants regardless of existing measurable disease as well.
Part 4 (expanded trial part): Overall Survival (OS) | From date of the first administration of 177Lu-PSMA-617 until date of death from any cause, assessed up to 2 years
  Overall survival (OS) is defined as the time (in months) from the date of the first administration of 177Lu-PSMA-617 to the date of death due to any cause. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive (on or before the cut-off date).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Japan (8):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Kyoto

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Takano S, Inaki A, Hirata K, Sparks RB, Sato M, Nomura S, Hattori T, Kambara H, Nguyen Q, Shiga T, Kinuya S, Hosono M. Pharmacokinetics and dosimetry of [177Lu]Lu-PSMA-617 and [68Ga]Ga-PSMA-11 in Japanese patients with PSMA-positive mCRPC. Ann Nucl Med. 2025 Nov;39(11):1201-1212. doi: 10.1007/s12149-025-02079-8. Epub 2025 Jul 10. PMID 40638023